CLINICAL TRIAL: NCT01151904
Title: Study of Brimonidine and Timolol Ophthalmic Solution With Latanoprost Compared With Latanoprost in Glaucoma Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty with patient recruitment
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-COM004
Record Dates: First submitted 2010-06-05; First posted 2010-06-29 (Estimated); Results first posted 2013-02-06 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-01

CONDITIONS: Glaucoma, Angle-Closure
MeSH Terms: conditions — Glaucoma, Angle-Closure | interventions — Brimonidine Tartrate; Timolol; Brimonidine Tartrate, Timolol Maleate Drug Combination; Latanoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- COMBIGAN® with Latanoprost (Experimental): Patients on current latanoprost monotherapy that qualify for study entry will have COMBIGAN® (brimonidine 0.2%/timolol 0.5% fixed combination ophthalmic solution) added to the latanoprost for 12 additional weeks.
  Interventions: Drug: brimonidine 0.2%/timolol 0.5% fixed combination ophthalmic solution; Drug: latanoprost

INTERVENTIONS:
Drug: brimonidine 0.2%/timolol 0.5% fixed combination ophthalmic solution — COMBIGAN® (brimonidine 0.2%/timolol 0.5% fixed combination ophthalmic solution) administered as one drop in the morning and one drop in the evening in affected eye(s) for 12 weeks.
  Other Names: COMBIGAN®
Drug: latanoprost — Latanoprost administered in the affected eye(s) as prescribed by physician.

SUMMARY:
This study will evaluate the safety and efficacy of patients switched from latanoprost monotherapy to a combination therapy of latanoprost with COMBIGAN® (brimonidine 0.2%/timolol 0.5% fixed combination ophthalmic solution) for chronic angle closure glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been administering latanoprost eye drops in affected eye(s) for at least 12 weeks prior to study
* Patient must have at least partially responded to latanoprost and requiring further IOP lowering eye drops
* Diagnosis of chronic angle-closure glaucoma
* Patients using COMBIGAN® in the past must not have been discontinued due to adverse events or lack of efficacy.

Exclusion Criteria:

* Known allergy or hypersensitivity to COMBIGAN®
* Corneal abnormalities that would preclude accurate IOP readings
* Any other active ocular disease other than glaucoma or ocular hypertension
* Ocular surgery within the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to lack of enrollment, this study was discontinued early.
Period: Overall Study
Arm/Group | COMBIGAN® With Latanoprost
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | COMBIGAN® With Latanoprost
Number analyzed (Participants) | 17
Age, Customized [Number; unit: Participants]
  <45 years | 0
  Between 45 and 65 years | 7
  >65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Intraocular Pressure (IOP)
Description: IOP is a measure of the fluid pressure inside the eye. A negative number change from baseline indicates a reduction in IOP (improvement). Due to lack of enrollment, analysis was not performed for this outcome measure.
Time Frame: Baseline, Week 12
Population: Planned analysis population: Intent to Treat: All enrolled patients who received at least 1 dose of study medication, had a valid baseline measurement, and at least one valid post-Day 0 IOP measure. Due to lack of enrollment, analysis was not performed for this outcome measure.
Arm/Group | COMBIGAN® With Latanoprost
Number analyzed (Participants) | 0

2. Secondary Outcome: Change From Baseline in IOP
Description: as for outcome 1
Time Frame: Baseline, Week 2, Week 6
Population: as for outcome 1
Arm/Group | COMBIGAN® With Latanoprost
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Responders With an IOP Reduction ≥20% From Baseline
Description: IOP is a measure of the fluid pressure inside the eye. A responder is defined as a patient with a mean IOP reduction of at least 20% in the affected eye(s) from baseline. Due to lack of enrollment, analysis was not performed for this outcome measure.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Arm/Group | COMBIGAN® With Latanoprost
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | COMBIGAN® With Latanoprost
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 5/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | COMBIGAN® With Latanoprost (N=17)
Corneal Erosion (Eye disorders) | 2
Conjunctival Hyperemia (Eye disorders) | 2
Somnolent (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
Due to lack of enrollment, this study was discontinued early and the outcome measures were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.